CLINICAL TRIAL: NCT03399084
Title: An Open-label, Randomized, Parallel, Bioequivalence Study of 750 mg Intravenous Single Dose Ferric Carboxymaltose Versus Injectafer® (750 mg Iron/15 mL Colloidal Solution) in Adult Patients With Iron Deficiency Anemia
Brief Title: A Study Comparing Two Ferric Carboxymaltose Formulations in Patients With Iron Deficiency Anemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1637 FCM_1
Record Dates: First submitted 2017-12-05; First posted 2018-01-16 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Iron Deficiency Anemia
Keywords: Ferric carboxymaltose; Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia | interventions — ferric carboxymaltose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ferric carboxymaltose (test) (Experimental): Patients will receive a single dose of Ferric carboxymaltose
  Interventions: Drug: Ferric carboxymaltose
- Ferric carboxymaltose (reference) (Active Comparator): Patients will receive a single dose of Ferric carboxymaltose
  Interventions: Drug: Ferric carboxymaltose

INTERVENTIONS:
Drug: Ferric carboxymaltose — 750 mg/15 mL

SUMMARY:
This study will evaluate bioequivalence of two formulations of Ferric Carboxymaltose as measured by serum total iron, in adult patients with iron deficiency anemia.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients at least 18 - 65 years of age;
* Patients with a body mass index (BMI) between 18.5 - 35 and with a body weight of ≥50 kg - ≤130 kg;

Exclusion Criteria:

* Patients with known hypersensitivity to ferric carboxymaltose, excipients, or similar product
* Patients with chronic kidney disease who are on dialysis of any kind.
* If female, is pregnant or nursing.
* Patients with blood loss leading to hemodynamic instability
* Patients with recent parenteral iron within 3 months prior to screening.

Other inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Bioequivalence assessed by maximum serum concentration (Cmax)of serum total iron. | Up to 7 days
  Measured by Cmax - The maximum plasma concentration of iron
Bioequivalence assessed by area under the serum concentration-time curve (AUC) of serum total iron. | Up to 7 Days
  Plasma Pharmacokinetics (PK) of study medication: Area Under the Plasma Concentration-time Curve (AUC)

SECONDARY OUTCOMES:
Maximum serum concentration (Cmax) of serum transferrin-bound iron. | Up to 7 days
  Plasma Pharmacokinetics (PK): The maximum plasma concentration
Time of Cmax (Tmax) of serum total iron and transferrin-bound iron | Up to 7 Days
  Plasma Pharmacokinetics (PK): Time of Cmax (Tmax)
Area under the serum concentration-time curve (AUC) of serum transferrin-bound iron | Up to 7 Days
  Plasma Pharmacokinetics (PK): area under the serum concentration-time curve (AUC)
Apparent terminal rate constant of serum total iron and transferrin-bound iron | Up to 7 Days
  Plasma Pharmacokinetics (PK): Apparent terminal rate constant
Apparent terminal half-life of serum total iron and transferrin-bound iron | Up to 7 Days
  Plasma Pharmacokinetics (PK): Apparent terminal half-life
Systemic clearance (CL) of serum total iron and transferrin-bound iron after intravenous dosing | Up to 7 Days
  Plasma Pharmacokinetics (PK): Systemic clearance (CL)
Volume of distribution at steady state of serum total iron and transferrin-bound iron following intravenous dosing | Up to 7 Days
  Plasma Pharmacokinetics (PK): Volume of distribution at steady state Plasma Pharmacokinetics (PK): Volume of distribution at steady state (Vss)
Number of patients with adverse events as a measure of safety and tolerability | Up to 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Sandoz Sandoz, Study Director — Novartis Pharmaceuticals
Locations (1):
- Sandoz Investigative Site, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com